CLINICAL TRIAL: NCT06883266
Title: Transcranial Direct Current Stimulation (tDCS) to Improve Motor Function and Motor Fatigue in Parkinson's Patients
Brief Title: Transcranial Direct Current Stimulation for Motor Function and Fatigue in PD
Acronym: tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH tDCS-Motor-PD
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Parkinsons Disease (PD)
Keywords: Parkinsons Disease; tDCS; Motor Function; Motor Fatigue
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an experimental group (receives stimulation) or a sham group (is set up with tDCS, but no stimulation is received)
Who Masked: Participant, Care Provider
Masking Description: The participant and their care provider will be blinded as to which intervention is being used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive 2mA of anodal transcranial direct current stimulation (tDCS) for 20 minutes daily for 5 consecutive days.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Sham Group (Sham Comparator): The sham group will be connected to the anodal transcranial direct current stimulation device daily for 5 days. During the 20 minute sessions, the participant will only receive stimulation for a 30-second ramp up period, at which point the stimulation will be discontinued for the remainder of the time.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — 2 mA will be administered for 5 consecutive days for a duration of 20 minutes with electrode placement at the left dorsolateral prefrontal cortex.
  Arms: Experimental Group
Device: Sham (No Treatment) — For 30 seconds, the patient will experience a ramp up of the stimulation, after which point no stimulation will be transmitted for the remainder of the session. This will be administered for 5 consecutive days for a duration of 20 minutes with electrode placement at the left dorsolateral prefrontal cortex
  Arms: Sham Group

SUMMARY:
The investigators hypothesize that multi-session anodal tDCS (atDCS) of the left primary motor cortex (M1) will induce long-lasting effects in improving motor function and reducing motor fatigue and fatigability in PD patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the fastest growing and second most common neurodegenerative disease (after Alzheimer's disease) and affects approximately one million people in the United States. Impaired motor function is one of the cardinal features of PD. One of the diagnostic criteria for PD is bradykinesia (slowness of movement). In addition to bradykinesia, PD patients also suffer from increased motor fatigue and motor fatigability. In the body of fatigue research, the term "motor fatigue' usually refers to the general sensation of tiredness or of difficulty in initiating physical activity experienced over several days to weeks. This is often assessed by questionnaires completed by the subject. The term 'motor fatigability' refers to difficulty in maintaining physical activity at a desired level (Lou, 2009). This is often assessed quantitively in a laboratory setting. Motor impairments, motor fatigue, and motor fatigability affect quality of life in patients with Parkinson's disease.

Transcranial direct current stimulation (tDCS) is a noninvasive and safe brain stimulation technique that has been shown to be effective in improving motor function in subjects with Parkinson's disease. During tDCS, low-voltage, low amplitude current is passed through a pair of surface electrodes placed over the areas of brain of interest.

The specific aim of this study is to examine if atDCS to M1 at 2 milliamps (mA) for 20 minutes daily for 5 days will improve motor function and reduce motor fatigue and fatigability in PD patients. The study will examine if the effects may last for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD with at least two of the four diagnostic criteria for PD (tremor, rigidity, bradykinesia, and postural instability)
* Must be able to consent

Exclusion Criteria:

* Patients with dementia (MOCA < 21)
* PD treatment using deep brain stimulation (DBS)
* Diagnosis of psychosis
* Diagnosis of multiple sclerosis
* Diagnosis of stroke
* Diagnosis of chronic obstructive pulmonary disease (COPD)
* Diagnosis of congestive heart failure (CHF)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Finger and Toe-Tapping on KinesiaOne Device | 30 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  We will use the KinesiaOne measure the finger tapping and foot tapping for 15 seconds. It will repeat 3 times at 1 minute intervals. KinesiaOne is a light-weight device that can be attached to the Index finger or ankle. It measures the acceleration and deceleration of the finger or foot. The measurement is transmitted to the KinesiaOne tablet that allows further data processing.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | 8 minutes; pre-test during the second research visit.
  This is a tool used to screen for mild cognitive dysfunctions. It assesses different domains of cognition: attention, memory, language visuospatial skills, orientation, and calculations. It determines the cut-off for dementia.
The Multidimensional Fatigue Inventory (MFI) | 5 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  This is a 20-item self-report instrument that measures five dimensions of fatigue independently: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity.
Center for Epidemiological Studies Depression Scale (CES-D). | 5 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  This is a tool used to screen for symptoms of depression.
McGill Quality of Life (QOL) Scale | 1 minute; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  This is a single item tool to assess quality of life on all parts of life (physical, emotional, social, spiritual, and financial.
MDS-UPDRS Part II (patient self-report) | 10 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  This is a 20-item patient self-report questionnaire that assess the motor aspects of experiences of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Shin Lou, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Brain and Spine Center, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126